CLINICAL TRIAL: NCT03055559
Title: Oral Iron Repletion With Globifer Forte® After 12 Weeks of Treatment
Brief Title: Trial Protocol GlobiFer - Oral Iron Repletion
Acronym: TPG
Status: Completed | Type: Observational
Sponsor: Gedeon Richter Slovakia, s.r.o. (Other)
Responsible Party: Sponsor
Other Study IDs: Not identified
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Iron Deficiency
Keywords: Iron, Hemoglobin, Feritin, erytrocyty. transferin
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Globifer Forte
  Interventions: Dietary Supplement: Globifer Forte

INTERVENTIONS:
Dietary Supplement: Globifer Forte

SUMMARY:
The haemoglobin level of the patients with iron deficiency should be increased clinical relevant after 12 weeks treatment with GlobiFer Forte.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 ≤ 60 years of age
2. Signed written informed consent
3. Hb ≥ 8 ≤ 10g/dl for
4. Female

Exclusion Criteria:

1. History of acquired iron overload, known haemochromatosis or first relatives with haemochromatosis, and allergic disorders (asthma, eczema, and anaphylactic reactions).
2. Known hypersensitivity to oral iron preparations.
3. Diseases, which an iron supplementation is not allowed or contraindicated.
4. Patients on current oral or intravenous iron supplementation
5. History of erythropoietin therapy in previous 30 days or scheduled for erythropoietin therapy or blood transfusion during duration of the study.
6. Patients who have had iron supplementation within the last 30 days.
7. Other reasons which in the investigator's judgment argue against inclusion of the patient into the trial.
8. Inability to comprehend study protocol
9. Participation in another clinical trial (currently or within the last 30 days)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female , ≥ 18 ≤ 60 years of age
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a clinical relevant increase of the haemoglobin level treatment with GlobiFer Forte | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ján Danko, PhD., Principal Investigator — Comenius University's Jessenius Faculty of Medicine
Locations (1):
- Prof. MUDr. Ján Danko, PhD., Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No